CLINICAL TRIAL: NCT02264522
Title: Use of Pulse Oximeter Derived Photo-plethysmographic Waveform to Guide Ultrafiltration in Hemodialysis Patients to Achieve Euvolemia While Minimizing Intra-dialytic Hypotension
Brief Title: Pilot Study Using a Pulse Oximeter Derived Photo-plethysmographic Waveform to Guide Hemodialysis Ultrafiltration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Intelomed, Inc. (Industry)
Collaborators: Centers for Dialysis Care, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 04-14-39
Record Dates: First submitted 2014-09-22; First posted 2014-10-15 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2016-08

CONDITIONS: Intradialytic Hypotension; Hypervolemia
MeSH Terms: conditions — Edema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm (Experimental): All patients will be enrolled in the same intervention arm. Interventions are implemented based in 1-4 event levels on the device. Interventions include: "Place dialysis chair into position 3", "Decrease dialysate temperature", "Decrease ultrafiltration rate by 25%", and "Decrease ultrafiltration rate by 50%".
  Interventions: Other: Place dialysis chair into position 3.; Other: Decrease dialysate temperature.; Other: Decrease ultrafiltration rate by 25%.; Other: Decrease ultrafiltration rate by 50%.

INTERVENTIONS:
Other: Place dialysis chair into position 3. — Upon device notification event 1, place patient in dialysis chair position 3.
Other: Decrease dialysate temperature. — Upon device notification event 2, decrease dialysate temperature by 0.5 degree centigrade.
Other: Decrease ultrafiltration rate by 25%. — Upon device notification event 3, decrease ultrafiltration rate by 25% from baseline ultrafiltration rate.
Other: Decrease ultrafiltration rate by 50%. — Upon device notification event 4, decrease ultrafiltration rate by 50% from baseline ultrafiltration rate.

SUMMARY:
The purpose of this study is to use the photo-plethysmographic [PPG] waveform signal to guide the dialysis and ultrafiltration [UF] of chronic maintenance hemodialysis patients, and to further the investigators understanding of homeostasis in hemodialysis.

The investigators hypothesize that the signals generated from the PPG device along with traditional monitoring and nursing judgment, will allow experienced, oriented staff to anticipate hemodynamic instability, intervene to prevent or mitigate the intradialytic hypotention [IDH], forestalling the onset of non-facilitating compensatory reflexes that preclude the patient from achieving an appropriate post-dialysis weight consistent with euvolemia. Furthermore, it is hypothesized that the nephrologist and staff will be able to wean patients from anti-hypertensive medications and craft patient specific dialysis orders and UF profiles that achieve consistent, comfortable treatment to appropriate end points.

The study aims include:

Aim 1: To confirm the temporal sequence of PPG signals and changes in BP in routine hemodialysis.

Aim 2: To refine further the predictive algorithms of PPG, augmented with continuous cardiac event monitoring (pre-intra-post hemodialysis) Aim 3: To develop targeted interventions to reverse the cardiovascular stress indicated by the PPG and to maintain perfusion.

Aim 4: To develop care paths approved by the medical staff and primary care nephrologist allowing RNs to respond to signals from the PPG.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years
2. On dialysis > 6 months with a stable dialysis program
3. Consistent achievement of a spKt/V ≥ 1.2
4. HGB ≥ 10 gm% ± ESA support
5. Consistent failure to achieve a post weight ≤ dry weight + 0.5Kg
6. Able to give informed consent directly
7. Frequent hypotensive reactions (≥ 1 / treatment in 4 of last 8 treatments)

   * Symptoms of hypotension
   * Intervention administered because of IDH (saline, "turn downs, early termination, trendelenberg position)
   * Drop in BP irrespective of symptoms. SBP < 90 mmHG intra or post HD if pre SBP was > 110 mmHG; SBP < 85 mmHG or 15 mmHG drop from start if starting BP ≤ 110 mmHG.
   * Or judged by the nursing staff to be difficult to achieve dry weight.

Exclusion Criteria:

1. Dialysis Catheter Access that may interfere with continuous data collection, per PI determination. (Catheter access is a relative exclusion based on the history of catheter performance.)
2. Cognitive Impairment precluding cooperation, and consent
3. Restless or unlikely to wear the monitor head-band
4. Too unstable in the judgment of their nephrologist to be included in a study of this nature.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-09; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Difference between prescribed dry weight and actual measured weight at end of dialysis session. | 8 weeks
  Percent difference between prescribed dry weight and actual weight at end of dialysis session.

CONTACTS AND LOCATIONS:
Locations (1):
- Centers for Dialysis Care - East, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No